CLINICAL TRIAL: NCT03738397
Title: A Phase 3b Multicenter, Randomized, Double-Blind, Double-Dummy, Active Controlled Study Comparing the Safety and Efficacy of Upadacitinib to Dupilumab in Adult Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Compare Safety and Efficacy of Upadacitinib to Dupilumab in Adult Participants With Moderate to Severe Atopic Dermatitis
Acronym: Heads Up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-046; 2018-002264-57 (EudraCT Number)
Expanded Access: NCT04159597 (Available)
Record Dates: First submitted 2018-11-09; First posted 2018-11-13 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Atopic Dermatitis
Keywords: Upadacitinib; ABT-494; Dupilumab; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib; dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Upadacitinib 30 mg QD (Experimental): Participants will receive 30 mg upadacitinib orally once a day (QD) up to Week 24 and placebo to dupilumab by subcutaneous injection every other week from Baseline to Week 22.
  Interventions: Biological: Upadacitinib; Drug: Placebo to dupilumab
- Dupilumab 300 mg EOW (Experimental): Participants will receive a loading dose of 600 mg dupilumab by subcutaneous (SC) injection on Day 1 followed by 300 mg dupilumab SC every other week (EOW) until Week 22 and placebo to upadacitinib orally QD up to Week 24.
  Interventions: Biological: Dupilumab; Drug: Placebo to upadacitinib

INTERVENTIONS:
Biological: Upadacitinib — Extended release tablet
  Other Names: ABT-494; RINVOQ®
  Arms: Upadacitinib 30 mg QD
Biological: Dupilumab — Dupilumab is administered as a subcutaneous (SC) injection
  Other Names: Dupixent®
  Arms: Dupilumab 300 mg EOW
Drug: Placebo to dupilumab — Placebo administered as a subcutaneous injection
  Arms: Upadacitinib 30 mg QD
Drug: Placebo to upadacitinib — Tablet
  Arms: Dupilumab 300 mg EOW

SUMMARY:
This study will evaluate upadacitinib compared to dupilumab (Dupixent®) in adults with moderate to severe atopic dermatitis (AD) who are candidates for systemic therapy.

DETAILED DESCRIPTION:
The study is comprised of a 35-day screening period, a 24-week double-blinded treatment period, and a follow-up visit 12 weeks after the last dose. Participants who complete Week 24 have the option to enroll into an open-label study (Study M19-850; NCT04195698) of upadacitinib 30 mg once daily and receive treatment with upadacitinib for an additional 52 weeks.

Participants who meet eligibility criteria will be randomized in a 1:1 ratio to receive either upadacitinib or dupilumab. Randomization will be stratified by Baseline disease severity (Validated Investigator Global Assessment scale for Atopic Dermatitis [vIGA-AD] score of moderate [3] versus severe [4]) and age (<40, ≥ 40 to < 65, ≥ 65 years).

ELIGIBILITY:
Inclusion Criteria:

* Participant has active moderate to severe atopic dermatitis (AD) defined by Eczema Area and Severity Index (EASI) ≥ 16, Investigator's Global Assessment (IGA) ≥ 3, ≥ 10% body surface area (BSA) of AD involvement at the Screening and Baseline Visits, and Baseline weekly average of daily Worst Pruritus NRS ≥ 4.
* Participant is a candidate for systemic therapy or have recently required systemic therapy for AD.

Exclusion Criteria:

* Participant has prior exposure to Janus Kinase (JAK) inhibitor.
* Participant has prior exposure to dupilumab.
* Participant is unable or unwilling to discontinue current AD treatments prior to the study.
* Participant has requirement of prohibited medications during the study.
* Participant has other active skin diseases or skin infections requiring systemic treatment or would interfere with appropriate assessment of AD lesions.
* Female participant who is pregnant, breastfeeding, or considering pregnancy during the study.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (159):
- United States (52):
  - Clinical Research Center AL /ID# 210277, Birmingham, Alabama
  - University of Arkansas for Medical Sciences /ID# 211688, Little Rock, Arkansas
  - Tien Q Nguyen MD, Inc /ID# 208934, Fountain Valley, California
  - UCSF Fresno /ID# 213253, Fresno, California
  - Jonathan Corren, MD. INC /ID# 208987, Los Angeles, California
  - California Allergy and Asthma Medical Group /ID# 213680, Los Angeles, California
  - Dermatology Research Associates /ID# 209097, Los Angeles, California
  - Los Angelos Cataract Center /ID# 208524, Los Angeles, California
  - Dermatology Clinical Trials /ID# 214622, Newport Beach, California
  - UC Davis Health /ID# 209285, Sacramento, California
  - Ucsd /Id# 208990, San Diego, California
  - Clinical Science Institute /ID# 211022, Santa Monica, California
  - The Community Research of South Florida /ID# 211145, Hialeah, Florida
  - Miami Dermatology and Laser Institute /ID# 212938, Miami, Florida
  - Florida International Rsrch cr /ID# 211562, Miami, Florida
  - Progressive Medical Research /ID# 211994, Port Orange, Florida
  - GCP Research /ID# 216020, St. Petersburg, Florida
  - Clinical Research Trials of Florida, Inc. /ID# 210751, Tampa, Florida
  - Integrated Clinical Research LLC /ID# 208831, West Palm Beach, Florida
  - Georgia Pollens Clinical Research Centers, Inc /ID# 211092, Albany, Georgia
  - Meridian Clinical Research Dermatology /ID# 213251, Savannah, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 208680, Chicago, Illinois
  - Medical Dermatology Associates of Chicago /ID# 210265, Chicago, Illinois
  - Sneeze, Wheeze, & Itch Associates, LLC /ID# 212058, Normal, Illinois
  - Dawes Fretzin, LLC /ID# 209187, Indianapolis, Indiana
  - Beacon Clinical Research, LLC /ID# 209280, Quincy, Massachusetts
  - Clarkston Skin Research /ID# 208739, Clarkston, Michigan
  - Henry Ford Health System /ID# 208741, Detroit, Michigan
  - Clinical Research Institute, Inc /ID# 210852, Minneapolis, Minnesota
  - Allergy, Asthma & Immunology Associates, PC /ID# 213481, Lincoln, Nebraska
  - Skin Specialists, PC /ID# 208843, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center /ID# 213727, Lebanon, New Hampshire
  - Forest Hills Dermatology Group /ID# 209249, Kew Gardens, New York
  - Montefiore Medical Center /ID# 209647, The Bronx, New York
  - Wake Forest Univ HS /ID# 208892, Winston-Salem, North Carolina
  - Univ Hosp Cleveland /ID# 208852, Cleveland, Ohio
  - The Ohio State University /ID# 209254, Columbus, Ohio
  - Southside Dermatology /ID# 212004, Tulsa, Oklahoma
  - Oregon Medical Res Center PC /ID# 208807, Portland, Oregon
  - Oregon Health and Science University /ID# 208809, Portland, Oregon
  - Medical University of South Carolina /ID# 211054, Charleston, South Carolina
  - Clinical Research Solutions, LLC /ID# 212542, Jackson, Tennessee
  - Orion Clinical Research /ID# 208765, Austin, Texas
  - DiscoveResearch, Inc. /ID# 213171, Bryan, Texas
  - Epiphany Dermatology - Fort Worth /ID# 211187, Fort Worth, Texas
  - Sante Clinical Research /ID# 212970, Kerrville, Texas
  - Stephen Miller, MD PA /ID# 210071, San Antonio, Texas
  - Sugar Land Allergy, Asthma, and Immunology Center /ID# 211153, Sugar Land, Texas
  - University of Utah /ID# 209001, Salt Lake City, Utah
  - Clinical Research Partners, LLC /ID# 212262, Richmond, Virginia
  - Premier Clinical Research /ID# 212142, Spokane, Washington
  - West Virginia Research Inst /ID# 212730, South Charleston, West Virginia
- Australia (5):
  - Holdsworth House Medical Practice /ID# 214565, Darlinghurst, New South Wales
  - The Skin Hospital /ID# 214401, Darlinghurst, New South Wales
  - Veracity Clinical Research /ID# 211134, Woolloongabba, Queensland
  - Sinclair Dermatology /ID# 209395, East Melbourne, Victoria
  - Burswood Dermatology /ID# 214875, Victoria Park, Western Australia
- Canada (10):
  - Kirk Barber Research, CA /ID# 209504, Calgary, Alberta
  - Dermatology Research Institute Inc. /ID# 210942, Calgary, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 211032, Surrey, British Columbia
  - Enverus Medical Research /ID# 209503, Surrey, British Columbia
  - Dr. Wei Jing Loo Medicine Prof /ID# 211400, London, Ontario
  - Lynderm Research Inc. /ID# 209505, Markham, Ontario
  - DermEdge Research Inc. /ID# 211122, Mississauga, Ontario
  - Niakosari Medicine Professional Corporation /ID# 211401, Toronto, Ontario
  - K. Papp Clinical Research /ID# 209509, Waterloo, Ontario
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 209498, Saint-Jérôme, Quebec
- Croatia (4):
  - DermaPlus - Poliklinika za dermatologiju i venerologiju /ID# 209935, Zagreb, City of Zagreb
  - Djecja bolnica Srebrnjak /ID# 209939, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 209976, Zagreb, City of Zagreb
  - Naftalan - Specijalna bolnica za medicinsku rehabilitaciju /ID# 209937, Ivanić-Grad, Zagreb County
- Czechia (5):
  - Fakultni Nemocnice Brno /ID# 212968, Brno
  - FN Hradec Kralove /ID# 209116, Hradec Králové
  - Nemocnice Jihlava, prispevkova organizace /ID# 209131, Jihlava
  - Fakultni nemocnice Ostrava /ID# 209117, Ostrava
  - Fakultni Nemocnice v Motole /ID# 209209, Prague
- Finland (4):
  - Keski-pohjanmaa Central Hospital /ID# 209534, Kokkola, Keski-Pohjanmaa
  - Oulu University Hospital /ID# 208961, Oulu, North Ostrobothnia
  - Mikkeli Central Hospital /ID# 210125, Mikkeli
  - Pihlajalinna Turku /ID# 209599, Turku
- France (7):
  - CHRU Lille - Hopital Claude Huriez /ID# 209317, Lille, Hauts-de-France
  - CHU de Nantes - Hotel Dieu /ID# 208974, Nantes, Pays de la Loire Region
  - Charles Nicolle CHU Rouen /ID# 208973, Rouen, Seine-Maritime
  - Hopital de la Timone /ID# 211245, Marseille
  - Centre Hospitalier Universitaire de Nice - Hopital l'Archet 2 /ID# 213374, Nice
  - Polyclinique Courlancy /ID# 208975, Reims
  - Hopital Larrey - CHU de Toulouse /ID# 208976, Toulouse
- Germany (6):
  - Universitatsklinikum Munster /ID# 210935, Munster, Lower Saxony
  - Gemeinschaftspraxis /ID# 211174, Blankenfeld-mahlow
  - Hautklinik Klinikum Darmstadt /ID# 210938, Darmstadt
  - Universitaetsklinikum Frankfurt /ID# 210934, Frankfurt
  - Medizinische Hochschule Hannover /ID# 210939, Hanover
  - TU Uniklinik Munchen /ID# 210937, Munich
- Hungary (5):
  - Oroshazi Korhaz /ID# 210150, Orosháza, Bekes County
  - Uno Medical Trials Kft /ID# 211177, Budapest XIII
  - Debreceni Egyetem Klinikai Kozpont /ID# 210893, Debrecen
  - Somogy Megyei Kaposi Mor Oktat /ID# 210149, Kaposvár
  - Pecsi Tudomanyegyetem Klinikai l.sz. Belgyogyaszati Klinika /ID# 210892, Pécs
- Ireland (2):
  - St Vincent's University Hosp /ID# 208441, Dublin
  - University Hospital Waterford /ID# 208442, Waterford
- Israel (4):
  - HaEmek Medical Center /ID# 210153, Afula
  - Rabin Medical Center /ID# 210012, Petah Tikva
  - Sheba Medical Center /ID# 210013, Ramat Gan
  - Ichilov Medical Center /ID# 210014, Tel Aviv
- Italy (7):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 210632, Milan, Lombardy
  - IBD Center - IRCCS Istituto Clinico Humanitas /ID# 215726, Rozzano, Milano
  - A.O. Policlinico Sant'Orsola Malpighi /ID# 209111, Bologna
  - A.O.U. di Brescia /ID# 209115, Brescia
  - Ospedale San Giovanni di Dio /ID# 209109, Cagliari
  - AO Univ di Modena /ID# 209110, Modena
  - Policlinico Univ Tor Vergata /ID# 209112, Rome
- Malaysia (6):
  - Hospital Sultan Ismail /ID# 211037, Johor Bahru, Johor
  - Hospital Pakar Sultanah Fatimah /ID# 210185, Muar town, Johor
  - UKM Medical Centre /ID# 209178, Kuala Lumpur, Selangor
  - Hospital Pulau Pinang /ID# 210212, George Town
  - University Malaya Med Ctr /ID# 208861, Kuala Lumpur
  - Hospital Putrajaya /ID# 209177, Putrajaya
- Netherlands (6):
  - Bravis Ziekenhuis /ID# 208584, Bergen op Zoom, North Brabant
  - Academisch Medisch Centrum /ID# 208578, Amsterdam, North Holland
  - Centrum Oosterwal /ID# 209641, Alkmaar
  - Universitair Medisch Centrum Groningen /ID# 208583, Groningen
  - Erasmus Medisch Centrum /ID# 208582, Rotterdam
  - Universitair Medisch Centrum Utrecht /ID# 208579, Utrecht
- New Zealand (3):
  - Optimal Clinical Trials Ltd /ID# 209475, Auckland
  - Clinical Trials NZ /ID# 215590, Hamilton
  - Wellington Hospital (Capital and Coast District Health Board) /ID# 215001, Wellington
- Norway (3):
  - St. Olavs Hospital HF /ID# 209137, Trondheim, Sor-Trondelag
  - Universitetssykehuset N-Norge, Harstad /ID# 209105, Harstad, Troms
  - Universitetssykehuset N-Norge, Tromso /ID# 209103, Tromsø, Troms
- Poland (6):
  - Szpital Uniwersytecki nr 1 im. dr. A. Jurasza w Bydgoszczy /ID# 211103, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Pratia MCM Krakow /ID# 207444, Krakow, Lesser Poland Voivodeship
  - Klinika Ambroziak Sp. z o.o. /ID# 207443, Warsaw, Masovian Voivodeship
  - Royalderm Agnieszka Nawrocka /ID# 211015, Warsaw, Masovian Voivodeship
  - ClinicMed Daniluk, Nowak Sp.j. /ID# 211112, Bialystok, Podlaskie Voivodeship
  - Dermoklinika Medical Center /ID# 211026, Lodz, Łódź Voivodeship
- Singapore (3):
  - National Skin Centre /ID# 208775, Singapore, Central Singapore
  - National University Hospital /ID# 208774, Singapore
  - Singapore General Hospital /ID# 208776, Singapore
- Spain (6):
  - Hospital Universitario de Bellvitge /ID# 207063, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Dr. Negrin /ID# 208969, Las Palmas de Gran Canaria, Las Palmas
  - Hospital de Manises /ID# 207062, Manises, Valencia
  - Complejo Hospitalario Universitario de Pontevedra /ID# 207139, Pontevedra
  - Hospital Universitario Arnau Vilanova /ID# 207065, Valencia
  - Hospital Universitario y Politecnico La Fe /ID# 207064, Valencia
- Sweden (2):
  - Skanes Universitetssjukhus /ID# 206783, Malmo, Skåne County
  - Karolinska University Hospital /ID# 207909, Stockholm
- Taiwan (4):
  - China Medical University Hosp /ID# 209770, Taichung, Taichung
  - National Taiwan University Hospital /ID# 208309, Taipei City, Taipei
  - Chung Shan Medical University /ID# 208311, Taichung
  - Taipei Municipal Wan Fang Hospital /ID# 209987, Taipei
- Ukraine (3):
  - Military Hospital of Military-Medical Clinical Center of Southern Region /ID# 210435, Zaporizhzhya, Zaporizhzhia Oblast
  - Kyiv City Clinical Skin and Venereal Hospital /ID# 210755, Kyiv
  - ME "Rivne Regional Dermatology and Venereology Dispensary" of RRC /ID# 210434, Rivne
- United Kingdom (6):
  - Royal Alex Childrens County Hospital /ID# 209709, Brighton, Brighton And Hove
  - Victoria Hospital /ID# 209853, Kirkcaldy, Fife
  - Royal Hospital for Children /ID# 210451, Glasgow, Glasgow City
  - The Royal Free Hospital /ID# 208659, London, London, City of
  - Guy's and St Thomas' NHS Found /ID# 208881, London, London, City of
  - Cardiff & Vale University Health Board /ID# 209745, Cardiff, Wales

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Result] Blauvelt A, Teixeira HD, Simpson EL, Costanzo A, De Bruin-Weller M, Barbarot S, Prajapati VH, Lio P, Hu X, Wu T, Liu J, Ladizinski B, Chu AD, Eyerich K. Efficacy and Safety of Upadacitinib vs Dupilumab in Adults With Moderate-to-Severe Atopic Dermatitis: A Randomized Clinical Trial. JAMA Dermatol. 2021 Sep 1;157(9):1047-1055. doi: 10.1001/jamadermatol.2021.3023. PMID 34347860
- [Derived] Simpson EL, Silverberg JI, Prajapati VH, Eyerich K, Katoh N, Boguniewicz M, Guttman-Yassky E, Song EJ, Lee WJ, Teixeira HD, Wu T, Sancho Sanchez C, Vigna N, Calimlim BM, de Bruin-Weller M. Rapid Itch Improvement and Skin Clearance with Upadacitinib Versus Placebo (Measure Up 1 and Measure Up 2) and Versus Dupilumab (Heads Up): Results from Three Phase 3 Clinical Trials in Patients with Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2025 Aug;15(8):2061-2076. doi: 10.1007/s13555-025-01443-w. Epub 2025 Jun 2. PMID 40457140
- [Derived] Blauvelt A, Eyerich K, Irvine AD, de Bruin-Weller M, Kwatra SG, Gooderham M, Kim B, Calimlim BM, Lee WJ, Raymundo EM, Liu Y, Ofori S, Platt AM, Silverberg JI. More Time Spent with Clear Skin and No Itch with Upadacitinib versus Dupilumab for Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Sep;14(9):2621-2630. doi: 10.1007/s13555-024-01242-9. Epub 2024 Aug 7. PMID 39110139
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 128 sites located in 22 countries (Australia, Canada, Croatia, Czechia, Finland, France, Germany, Hungary, Ireland, Israel, Italy, Malaysia, Netherlands, New Zealand, Norway, Poland, Singapore, Spain, Taiwan, Ukraine, United Kingdom, and the United States).
Pre-assignment Details: Participants were randomly assigned in a 1:1 ratio to receive upadacitinib or dupilumab. Randomization was stratified by disease severity (Validated Investigator Global Assessment Scale for Atopic Dermatitis [vIGA-AD] moderate [3] vs severe [4]) and age (<40, ≥ 40 to < 65, ≥ 65 years).
Groups:
- Dupilumab 300 mg EOW: Participants received a loading dose of 600 mg dupilumab by subcutaneous (SC) injection on Day 1 followed by 300 mg dupilumab SC every other week (EOW) until Week 22 and placebo to upadacitinib orally once a day (QD) up to Week 24.
- Upadacitinib 30 mg QD: Participants received 30 mg upadacitinib orally once a day up to Week 24 and placebo to dupilumab SC EOW up to Week 22.
Period: Overall Study
Arm/Group | Dupilumab 300 mg EOW | Upadacitinib 30 mg QD
Started | 331 | 342
Completed | 308 | 312
Not Completed | 23 | 30
Not completed — Adverse Event | 3 | 7
Not completed — Withdrawal by Subject | 8 | 11
Not completed — Lost to Follow-up | 7 | 5
Not completed — COVID-19 Logistical Restrictions | 1 | 1
Not completed — Other | 4 | 6

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population includes all randomized participants according to the treatment groups that they were randomized to.
Groups:
- Dupilumab 300 mg EOW: Participants received a loading dose of 600 mg dupilumab by SC injection on Day 1 followed by 300 mg dupilumab SC EOW until Week 22 and placebo to upadacitinib orally QD up to Week 24.
- Total: Total of all reporting groups
Arm/Group | Dupilumab 300 mg EOW | Upadacitinib 30 mg QD | Total
Number analyzed (Participants) | 331 | 342 | 673
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (13.81) | 36.2 (14.42) | 36.3 (14.11)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 223 | 228 | 451
  ≥ 40 to < 65 years | 94 | 98 | 192
  ≥ 65 years | 14 | 16 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 159 | 298
  Male | 192 | 183 | 375
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 25 | 56
  Not Hispanic or Latino | 300 | 317 | 617
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 231 | 229 | 460
  Black or African American | 15 | 25 | 40
  Asian | 78 | 77 | 155
  American Indian/Alaska Native | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Multiple | 5 | 6 | 11
Disease Severity [Count of Participants; unit: Participants] — Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) was used to assess the severity of AD based on lesion appearance on the following scale:
  * 0-Clear: No signs of AD;
  * 1-Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2-Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  * 3-Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, possible oozing or crusting;
  * 4-Severe: Marked erythema, induration/papulation and/or lichenification.
  Participants
    3 (Moderate) | 159 | 169 | 328
    4 (Severe) | 172 | 173 | 345
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: score on a scale] — EASI is a tool to measure the extent and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected, and the severity of eczema (scored as none [0], mild [1], moderate [2], or severe [3]) for redness, thickness, scratching, and lichenification are assessed. The EASI score is the sum of the scores for each region and ranges from 0 to 72, where higher scores represent worse disease.
  score on a scale | 29.21 (11.551) | 30.96 (12.550) | 30.10 (12.092)
Duration Since AD Diagnosis [Mean (Standard Deviation); unit: years] | 25.474 (14.8251) | 23.608 (14.7697) | 24.526 (14.8154)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a 75% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 75) at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population; non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab 300 mg EOW | Upadacitinib 30 mg QD
Number analyzed (Participants) | 331 | 342
percentage of participants | 62.6 [57.4 to 67.8] | 72.4 [67.6 to 77.2]
Statistical Analysis 1: Comparison: Dupilumab 300 mg EOW vs Upadacitinib 30 mg QD; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel — A multiple testing procedure was used to provide a strong control of the type I error rate at alpha = 0.05 (2-sided) across analyses comparing upadacitinib versus dupilumab with respect to the primary and ranked secondary endpoints; Cochran-Mantel-Haenszel test adjusted for vIGA-AD categories (moderate [3] versus severe [4]); Adjusted Response Rate Difference = 9.7, 95% CI 2-sided [2.6 to 16.7] — Response rate difference = Upadacitinib - Dupilumab

2. Secondary Outcome: Percent Change From Baseline in Worst Pruritus Numerical Rating Scale (NRS) Score at Week 16
Description: The Worst Pruritus NRS is an assessment tool that participants used to report the intensity of their pruritus during a 24-hour recall period using an electronic hand-held device. Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
  The percent change from Baseline was calculated from a rolling weekly average; a negative change from Baseline indicates improvement.
Time Frame: Baseline (Week 0) to Week 16
Population: Intent-to-treat population with non-missing Baseline and at least one post-baseline value; missing data were handled using a mixed-effect model with repeated measurements (MMRM) including observed measurements at all visits, except that measurements after any rescue medication were excluded.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Dupilumab 300 mg EOW | Upadacitinib 30 mg QD
Number analyzed (Participants) | 239 | 252
percent change | -49.58 (1.986) | -67.78 (1.906)
Statistical Analysis 1: Comparison: Dupilumab 300 mg EOW vs Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; Mixed-effect model repeat measurement with Baseline, treatment, visit, treatment by visit interaction, and Baseline vIGA-AD categories in the model; Least Squares (LS) Mean Difference = -18.21, 95% CI 2-sided [-23.61 to -12.80], Standard Error of Mean 2.753 — Difference = Upadacitinib - Dupilumab

3. Secondary Outcome: Percentage of Participants Achieving a 100% Reduction From Baseline in EASI Score (EASI 100) at Week 16
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab 300 mg EOW | Upadacitinib 30 mg QD
Number analyzed (Participants) | 331 | 342
percentage of participants | 7.9 [5.0 to 10.8] | 28.4 [23.6 to 33.2]
Statistical Analysis 1: Comparison: Dupilumab 300 mg EOW vs Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel test adjusted for vIGA-AD categories (moderate [3] versus severe [4]); Adjusted Response Rate Difference = 20.4, 95% CI 2-sided [14.8 to 26.0] — Response rate difference = Upadacitinib - Dupilumab

4. Secondary Outcome: Percentage of Participants Achieving a 90% Reduction From Baseline in EASI Score (EASI 90) at Week 16
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab 300 mg EOW | Upadacitinib 30 mg QD
Number analyzed (Participants) | 331 | 342
percentage of participants | 40.3 [35.0 to 45.6] | 61.6 [56.4 to 66.8]
Statistical Analysis 1: Comparison: Dupilumab 300 mg EOW vs Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel test adjusted for vIGA-AD categories (moderate [3] versus severe [4]); Adjusted Response Rate Difference = 21.2, 95% CI 2-sided [13.8 to 28.6] — Response rate difference = Upadacitinib - Dupilumab

5. Secondary Outcome: Percent Change From Baseline in Worst Pruritus Numerical Rating Scale (NRS) Score at Week 4
Description: as for outcome 2
Time Frame: Baseline (Week 0) to Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Dupilumab 300 mg EOW | Upadacitinib 30 mg QD
Number analyzed (Participants) | 297 | 327
percent change | -32.39 (2.288) | -60.41 (2.204)
Statistical Analysis 1: Comparison: Dupilumab 300 mg EOW vs Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -28.02, 95% CI 2-sided [-34.25 to -21.78], Standard Error of Mean 3.177 — Difference = Upadacitinib - Dupilumab

6. Secondary Outcome: Percentage of Participants Achieving a 75% Reduction From Baseline in EASI Score at Week 2
Description: as for outcome 1
Time Frame: Baseline and Week 2
Population: Intent-to-treat population; Non-responder imputation while incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab 300 mg EOW | Upadacitinib 30 mg QD
Number analyzed (Participants) | 331 | 342
percentage of participants | 18.2 [14.0 to 22.4] | 44.3 [39.1 to 49.6]
Statistical Analysis 1: Comparison: Dupilumab 300 mg EOW vs Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel test adjusted for vIGA-AD categories (moderate [3] versus severe [4]); Adjusted Response Rate Difference = 26.0, 95% CI 2-sided [19.3 to 32.7] — Response rate difference = Upadacitinib - Dupilumab

7. Secondary Outcome: Percent Change From Baseline in Worst Pruritus Numerical Rating Scale (NRS) Score at Week 1
Description: as for outcome 2
Time Frame: Baseline (Week 0) to Week 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Dupilumab 300 mg EOW | Upadacitinib 30 mg QD
Number analyzed (Participants) | 314 | 331
percent change | -8.94 (1.831) | -31.96 (1.772)
Statistical Analysis 1: Comparison: Dupilumab 300 mg EOW vs Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -23.02, 95% CI 2-sided [-28.03 to -18.02], Standard Error of Mean 2.548 — Difference = Upadacitinib - Dupilumab

8. Secondary Outcome: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 16
Description: The Worst Pruritus NRS is an assessment tool that participants used to report the intensity of their pruritus during a 24-hour recall period using an electronic hand-held device. Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
Time Frame: Baseline and Week 16
Population: Intent-to-treat population with Worst Pruritus NRS ≥ 4 at Baseline; non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab 300 mg EOW | Upadacitinib 30 mg QD
Number analyzed (Participants) | 323 | 334
percentage of participants | 36.4 [31.1 to 41.6] | 56.1 [50.8 to 61.5]
Statistical Analysis 1: Comparison: Dupilumab 300 mg EOW vs Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel test adjusted for vIGA-AD categories (moderate [3] versus severe [4]); Adjusted Response Rate Difference = 19.8, 95% CI 2-sided [12.4 to 27.3] — Response rate difference = Upadacitinib - Dupilumab

ADVERSE EVENTS:
Time Frame: All-cause mortality was recorded from Day 1 up to 12 weeks after last injection (34 weeks). Treatment-emergent adverse events are from first dose of upadacitinib/dupilumab through 30 days following the last dose of upadacitinib or 84 days following the last dose of dupilumab (up to 34 weeks).
Arm/Group | Dupilumab 300 mg EOW | Upadacitinib 30 mg QD
All-Cause Mortality (participants affected / at risk) | 0/331 | 1/342
Serious Adverse Events (participants affected / at risk) | 7/331 | 14/342
Other Adverse Events (participants affected / at risk) | 134/331 | 167/342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 300 mg EOW (N=331) | Upadacitinib 30 mg QD (N=342)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
GLAUCOMA (Eye disorders) | 0 (0) | 1 (1)
INCARCERATED UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
FOOD ALLERGY (Immune system disorders) | 0 (0) | 1 (1)
TYPE I HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
BETA HAEMOLYTIC STREPTOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
PELVIC ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INTENTIONAL SELF-INJURY (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ABORTION INDUCED (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 300 mg EOW (N=331) | Upadacitinib 30 mg QD (N=342)
CONJUNCTIVITIS (Infections and infestations) | 35 (36) | 5 (6)
FOLLICULITIS (Infections and infestations) | 4 (4) | 22 (22)
NASOPHARYNGITIS (Infections and infestations) | 27 (31) | 23 (33)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 17 (20) | 26 (26)
URINARY TRACT INFECTION (Infections and infestations) | 15 (16) | 18 (19)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 10 (12) | 26 (27)
HEADACHE (Nervous system disorders) | 24 (32) | 17 (22)
ACNE (Skin and subcutaneous tissue disorders) | 11 (12) | 64 (72)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 32 (51) | 36 (52)
ORAL HERPES (Infections and infestations) | 9 (10) | 17 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT03738397/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT03738397/SAP_001.pdf